CLINICAL TRIAL: NCT03193892
Title: A National Registry on Clinical Manifestations, Genetics, Interventions, and Outcomes in Chinese Patients With Lymphangioleiomyomatosis (LAM-CHINA)
Brief Title: A National Registry on Chinese Patients With Lymphangioleiomyomatosis
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Guangzhou Institute of Respiratory Disease (Other); Central South University (Other); Anhui Provincial Hospital (Other Government); Xiangya Hospital of Central South University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Wuxi People's Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); West China Hospital (Other); Fujian Provincial Hospital (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC091502LAM
Record Dates: First submitted 2017-06-14; First posted 2017-06-21 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Function
Keywords: registry; China; lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biological specimens are preserved in serum, plasma, and leukocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary lymphangioleiomyomatosis (LAM), a disease characterized by diffuse cystic changes in the lung, is a rare disorder that affects almost exclusively women. The main objectives of this study are to accurately evaluate the prevalence of LAM, the status of disease, the diagnosis and treatment, the quality of care, and the health related outcomes in China.

DETAILED DESCRIPTION:
Pulmonary lymphangioleiomyomatosis (LAM), a disease characterized by diffuse cystic changes in the lung, is a rare disorder that affects almost exclusively women. The main objectives of this study are to accurately evaluate the prevalence of LAM, the status of disease, the diagnosis and treatment, the quality of care, and the health related outcomes in China. This is a register study lasting 4 years, aims to raise 800 subjects. Primary endpoint is the annual change of forced expiratory volume in the first second (FEV1) and forced vital capacity (FVC) in pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: female.
2. Age: no limitation.
3. Diagnosis meets one of the following criteria, (1) definite or probable diagnosis of LAM based on ATS/JRS and ERS criteria. (2) Investigators recommend including of the patient.

Exclusion Criteria:

1. Suspected LAM patients without other supporting evidence for LAM diagnosis.
2. No diffuse cystic lesions in the lung.
3. Patients with bilateral cystic lung lesions but the LAM diagnosis cannot be established.
4. Without signed informed consent.
5. Difficult to follow up.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pulmonary lymphangioleiomyomatosis (LAM) affects almost exclusively women.
Study Population: Study Population is from across the country of China.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in spirometry (FEV1 and FVC) of lymphangioleiomyomatosis patients. | 10 years
  Spirometry will be evaluated at baseline and through study completion, an average of 3 years.

SECONDARY OUTCOMES:
Change of diffusing capacity of the lung. | 10 years
  Pulmonary function tests will be evaluated at baseline and through study completion, an average of 3 years.
Annual incidence of major health outcomes: hemoptysis, pneumothorax, chylothorax, and spontaneous hemorrhage of kidney angiomyolipoma (AML). | 10 years
  The number of occurrences will be recorded through study completion, an average of 3 years.
Other health outcomes: pregnancy, malignant tumors except LAM, lung transplantation, and death. | 10 year
  The number of occurrences will be recorded through study completion, an average of 3 years.
The incidence of adverse drug reactions of long-time treatment with rapamycin. | 10 years
  Common Terminology Criteria for Adverse Events (CTCAE) will be used to evaluate adverse drug reactions through study completion, an average of 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Currently, there is no such a plan to share IPD to other researchers

REFERENCES:
- [Derived] Wang YY, Zou LP, Xu KF, Xu WS, Zhang MN, Lu Q, Tian XL, Pang LY, He W, Wang QH, Gao Y, Liu LY, Chen XQ, Ma SF, Chen HM, Dun S, Yang XY, Luo XM, Huang LL, Li YF. Long-term safety and influence on growth in patients receiving sirolimus: a pooled analysis. Orphanet J Rare Dis. 2024 Aug 15;19(1):299. doi: 10.1186/s13023-024-03243-5. PMID 39148107
- [Derived] Xu W, Yang C, Cheng C, Wang Y, Hu D, Huang J, He Y, Wang J, Chen K, Yang L, Zhou W, Zhang T, Liu S, Dai J, Meng S, Li X, Yang Y, Wang ST, Feng R, Zhang W, Zhang H, Wang L, Tian X, Xu KF. Determinants of Progression and Mortality in Lymphangioleiomyomatosis. Chest. 2023 Jul;164(1):137-148. doi: 10.1016/j.chest.2023.02.026. Epub 2023 Feb 18. PMID 36801466